CLINICAL TRIAL: NCT07029204
Title: Pilot Study on Intralesional Cyclosporine for Alopecia Areata
Brief Title: Intralesional Cyclosporine for Alopecia Areata
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2168339
Record Dates: First submitted 2025-05-08; First posted 2025-06-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Cyclosporine; Intralesional Injection
MeSH Terms: conditions — Alopecia Areata | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Blinded Cyclosporine Injection (Experimental): Two lesions on each participant are chosen and randomized. One lesion will receive an intralesional injection of 0.5-2 mL of cyclosporine (2.5 mg/ml) depending on lesion size. The injection will be given weekly for 8 weeks.
  Interventions: Drug: CycloSPORINE Injectable Product
- Blinded Placebo Injection (Placebo Comparator): Two lesions on each participant are chosen and randomized. One lesion will receive an intralesional injection of 0.5-2 mL of saline solution depending on lesion size. The injection will be given weekly for 8 weeks.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: CycloSPORINE Injectable Product — Intralesional 0.5-2 mL injections of cyclosporine (2.5 mg/ml)
  Arms: Blinded Cyclosporine Injection
Drug: Saline Solution — Intralesional 0.5-2 mL injections of Saline Solution
  Arms: Blinded Placebo Injection

SUMMARY:
Alopecia areata (AA) is a chronic autoimmune disease that causes non-scarring, focal areas of hair loss. Due to its resulting disfigurement and unpredictable course, it is recognized as a serious medical condition with severe emotional and psychosocial distress, including a high prevalence of depression and anxiety.1-4 Treatment options for alopecia areata are limited.

Cyclosporine has been used as an effective therapeutic option in the treatment of psoriasis. Additionally, the use of oral cyclosporine, alone or in combination with other agents, has been used in the management of a multitude of dermatologic conditions, including alopecia areata, pyoderma gangrenosum, chronic idiopathic purpura, atopic dermatitis, dyshidrotic eczema, Behcet disease, dermatomyositis, among others.8

Although cyclosporine has demonstrated efficacy in the management of these diseases, systemic side effects of oral cyclosporine often limit its long-term use. However, intralesional injections of cyclosporine have not been investigated. Through this randomized double-blind placebo-controlled clinical study, the study team aims to evaluate the safety, dosing, and efficacy of intralesional cyclosporine for use in the treatment of alopecia areata. The study team expects about 12 people at UC Davis to take part in this research. The study itself includes 11 visits and will last about 12 weeks.

DETAILED DESCRIPTION:
Alopecia areata (AA) is a chronic autoimmune disease that causes non-scarring, focal areas of hair loss. Due to its resulting disfigurement and unpredictable course, it is recognized as a serious medical condition with severe emotional and psychosocial distress, including a high prevalence of depression and anxiety.1-4 Treatment options for alopecia areata are limited. Currently, baricitinib is the only FDA-approved treatment for alopecia areata. However, in clinical trials, only 39% of patients receiving the highest dose of baricitinib achieved the primary endpoint of a Severity of Alopecia Tool score of <20 at week 36, thus demonstrating a need for more efficacious therapies.5

Cyclosporine has been used as an effective therapeutic option in the treatment of psoriasis. Additionally, the use of oral cyclosporine, alone or in combination with other agents, has been used in the management of a multitude of dermatologic conditions, including alopecia areata, pyoderma gangrenosum, chronic idiopathic purpura, atopic dermatitis, dyshidrotic eczema, Behcet disease, dermatomyositis, among others.8

Although cyclosporine has demonstrated efficacy in the management of these diseases, particularly with severe and recalcitrant disease course, systemic side effects of oral cyclosporine often limit its long-term use. These risks include hypertension, nephrotoxicity, prolonged immunosuppression, hyperkalemia, and hypomagnesemia.9 In consideration of these systemic adverse effects, it is important to investigate alternatives mechanisms of drug administration, including intralesional injections, to facilitate more localized drug delivery while minimizing systemic toxicity.

Oral cyclosporine has been used in the treatment of alopecia areata as a steroid-sparing agent. However, intralesional injections of cyclosporine have not been investigated. Through this randomized double-blind placebo-controlled clinical study, the study team aims to evaluate the safety, dosing, and efficacy of intralesional cyclosporine for use in the treatment of alopecia areata.

The study team expects about 12 people at UC Davis to take part in this research. The study itself includes 11 visits and will last about 12 weeks. Each participant will be evaluated and two similar areas affected by alopecia areata will be selected. These two areas will be randomly assigned to either treatment or placebo. Both participants and investigators will be blinded to treatment assignments. The participant will receive the two weekly injections, a disease activity assessment, a physical examination, vital collection, standardized photography, and surveys during each visit in the treatment phase of the study. Blood work will be completed biweekly. After week 8, one follow up will be scheduled during week 12 where the participant will be assessed again.

Through conducting this study, the study team aims to collect preliminary insights regarding the safety, dosing, and efficacy of intralesional cyclosporine for alopecia areata, guiding future larger-scale investigations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 at screening visit.
* Diagnosis of alopecia areata by a board-certified dermatologist at screening visit.
* Current alopecia areata episode involving the scalp of more than 3 months' duration prior to baseline visit.
* SALT Score between 10 and 50 at baseline visit.
* Stable disease based on subject history over the past 1 month.
* Agree not to use any alopecia areata treatments during the study, including, but not limited to: systemic therapies (eg, methotrexate, cyclosporine, corticosteroids, JAK inhibitors) and biologics (eg, monoclonal antibodies), intralesional corticosteroid injections, topical therapies, and phototherapy

Exclusion Criteria:

* Currently experiencing other forms of alopecia. Including but not limited to: androgenetic alopecia, telogen effluvium, or any other concomitant conditions (eg, tinea capitis, psoriasis, lupus erythematosus, or secondary syphilis) that could interfere with evaluation of alopecia areata
* Previous treatment with cyclosporine
* Other autoimmune diseases
* Pregnancy or lactation
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking study drug or interfere with the interpretation of data. These may include, but are not limited to, patients with untreated hypertension, patients with known renal disease with decreased GFR, and known infection.
* Adults unable to consent
* Prisoners
* Currently using drugs that are well-substantiated to interact with cyclosporine, including the following: ciprofloxacin, gentamicin, tobramycin, trimethoprim with sulfamethaxazole, vancomycin, melphalan, amphotericin B, ketoconazole, azapropazon, colchicine, diclofenac, naproxen, sulindac, cimetidine, ranitidine, tacrolimus, fibric acid derivatives (e.g. bezafibrate, fenofibrate), and methotrexate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Hair Regrowth: SALT Score | Screening to Week 12
  Using the Severity of Alopecia Tool (SALT), study team will track and monitor the percentage of scalp hair loss throughout participant's duration in the trial.
Hair Regrowth: PRO for scalp hair assessment | Week 0 and Week 12
  PRO for scalp hair assessment will be a questionnaire given to participants where they will elevate their hair loss on a scale of 0-4.
Hair Regrowth: Standardized photographs | Week 0 to Week 12
  Standardized photographs of participant's scalps will be taken throughout the course of the study to visual monitor outcomes. There will be a minimum of 5 photographs taken: one of each of the 4 planes of scalp and 1 frontal view of face and scalp. These photographs will be compared to one another through the study to assess the hair regrowth that occurred following the cyclosporine injections.

SECONDARY OUTCOMES:
Safety End Point: Adverse Events | Screening to Week 12
  To assess any adverse events that may be associated with the study or its procedures
Liver Function: Alanine transaminase (ALT), Aspartate transaminase (AST), Alkaline phosphatase (ALP) measured in units per liter (U/L) | Week 0 to Week 12
  Blood samples will be used to evaluate ALT, AST, and ALP levels to determine if cyclosporine or study procedures may affect liver function.
Kidney Function: Blood Urea Nitrogen (BUN) and Creatinine measured in milligrams per deciliter (mg/dL) | Week 0 to Week 12
  Blood samples will be used to evaluate BUN and Creatinine levels to determine if cyclosporine or study procedures may affect kidney function.
Number of participants with abnormal Complete Blood Count (CBC) | Week 0 to Week 12
  Through patient blood samples, abnormalities in CBC will be noted and the total number of patients will be evaluated.
Cyclosporine levels measured in nanograms per milliliter (ng/mL) | Week 0 to Week 12
  Blood samples will be used to evaluate cyclosporine levels in blood due to intralesional cyclosporine injection.
Blood Pressure measured in millimeters of mercury (mm Hg) | Screening to Week 12
  Diastolic and Systolic blood pressure will be collected before and after intralesional injection throughout the study to assess if cyclosporine or study procedures may have an effect.
Heart Rate measured in beats per minute (b/m) | Screening to Week 12
  Heart rate will be measured using a vital machine before and after intralesional injection throughout the study to assess if cyclosporine or study procedures may have an effect.
Temperature measured in Fahrenheit (F) | Screening to Week 12
  Temperature will be measured using a thermometer before and after intralesional injection throughout the study to assess if cyclosporine or study procedures may have an effect.

CONTACTS AND LOCATIONS:
Overall Officials: Oma Agbai, MD, Principal Investigator — UC Davis Health Department of Dermatology
Locations (1):
- University of California, Davis - Dermatology Department, Sacramento, California, United States